CLINICAL TRIAL: NCT02583958
Title: Assessment of Efficacy and Safety for a New Wound Dressing URGO 310 3166 in the Local Treatment of Venous or Mixed Leg Ulcers: A European, Randomised Clinical Trial
Brief Title: Assessment of Efficacy & Safety for a New Wound Dressing Urgo 310 3166 in the Local Treatment of VLU or Mixed Leg Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FI-14-06-310 3166
Record Dates: First submitted 2015-10-12; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device Urgo 3103166 (Experimental): Soft-adherent hydro-desloughing dressing
  Interventions: Device: Urgo 3103166
- Device Aquacel Extra (Active Comparator): Hydrofibre dressing
  Interventions: Device: Aquacel Extra

INTERVENTIONS:
Device: Urgo 3103166 — URGO 310 3166 dressing should be changed as often as required (let to the Investigator's convenience). The dressing change frequency is based on the exudate level and the clinical progress of the wound (up to 7 days).
  Arms: Device Urgo 3103166
Device: Aquacel Extra — Aquacel Extra hydrofibre dressing can be left in place up to 7 days, where clinically indicated.
  Arms: Device Aquacel Extra

SUMMARY:
Assessment of efficacy and safety for a new wound dressing URGO 310 3166 in the local treatment of venous or mixed leg ulcers: a European, randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old who has provided his/her written informed consent,
* Patient who can be monitored by the same investigation team throughout the whole duration of the study,
* Patient who agrees to wear an effective venous compression system every day, associated with the trial dressing,
* Leg ulcer with an Ankle Brachial Pressure Index (ABPI) not less than 0.7 and not more than 1.3,
* Ulcer area > or equal to 5cm2,
* Ulcer duration > or equal to 6 months,
* Ulcer presenting a the surface wound bed covered with 50% or more by sloughy tissue,
* Moderately or heavily exudative ulcers.

Exclusion Criteria:

* Clinical infection on the wound bed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Relative regression of wound surface area | week 20

SECONDARY OUTCOMES:
Percentage of debrided wounds | at each clinical evaluation up to 20 weeks
Occurrence of adverse events as assessed by the investigator according to a classification MedDRA | between inclusion and week 20
Patient's Quality of Life | at inclusion visit and at week 20 or at the end of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Meaume, MD, Principal Investigator — Hospital Rothschild - Paris - France
Locations (1):
- Hospital Rothschild, Paris, France